CLINICAL TRIAL: NCT03558282
Title: Facial Mucosal Level Determinants for Single Immediately Placed Implants Evaluated by Novel Ultrasonography
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Kuwait Foundation for the Advancement of Sciences (Unknown)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Clinical Assistant Professor, University of Michigan
Other Study IDs: HUM00139630
Record Dates: First submitted 2018-05-18; First posted 2018-06-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maxillary Anterior Implant: Subjects who have a single implant restoration in the maxillary anterior position with sufficient baseline data. Recession observation and crown contour observation of the implant will be completed.
  Interventions: Other: Recession Observation; Diagnostic Test: Crown Contour Observation

INTERVENTIONS:
Other: Recession Observation — Soft tissue measurements
Diagnostic Test: Crown Contour Observation — Ultrasound measures of implant crown contour.

SUMMARY:
A single center, prospective clinical trial is planned to investigate the effect of different emergence angles of implant restorations on peri-implant soft tissue recession and implant marginal bone loss.

The primary outcome is to systematically evaluate the association of implant-, peri-implant tissue-, and restoration-related factors with facial mucosal level changes.

DETAILED DESCRIPTION:
Facial mucosal recession still poses a threat to long-term success of implant therapy especially esthetic appearance. To study the timing and extent of mucosal recession and the associated risks, a prospective study is strategically important. This will allow the collection of valuable longitudinal data about facial mucosal level changes, peri-implant tissue dimensions, and implant/restoration parameters that are considered critical for determining the mucosal level. Forty adult patients who meet the inclusion criteria will be recruited to participate in this study. Patients that had an implant crown placed a minimum time frame of 6 months and have existing relevant clinical data (mucosal level and thickness, radiographs, cone beam computed tomogram (CBCT) scans, study casts and intra-oral photographs) at baseline and if possible at other follow-up visits will be invited to participate in this study. Patients that volunteer to be screened will not be examined for study eligibility until an informed consent has been obtained. Patient information will be protected according to HIPAA. The enrolled subjects will have research measurements taken, an ultrasound scan, intraoral photos and an impression of the arch including the study implant. One dental cone beam computed tomography (CBCT) scan will be taken to evaluate the implant position in relation to the alveolar ridge and to evaluate relative bone quality. The primary outcome will analyze the changes in the facial mucosal level, by superimposing the digital images of the stone models that were taken previously. On ultrasound images, peri-implant tissue parameters, implant positions, restoration contour, etc., will be measured and recorded. The primary outcome will then be equated with clinical and radiographic readings, and ultrasound parameters, along with timing of provisionalization or final restoration, in regression analysis to identify factors related to facial mucosal recession.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years old or older
* One immediate maxillary implant placement with 2 adjacent neighboring teeth
* Available pre-surgery model
* Radiographic documentation (either peri-apical x-rays or CBCT)
* Have final restoration for at least 6 months.

Exclusion Criteria:

* Are under 18 years of age.
* Are unwilling or unable to read and sign this informed consent document.
* Have any medical conditions that we believe may influence the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who had a single implant restoration in the maxillary anterior position with sufficient baseline data will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Mucosal recession on the tested implant | At least 12 months following implant placement.
  It is a one-time measurement (this study is only one-time visit) within the study timeframe, measured from a reference, adjacent tooth landmark, to the mucosal margin of the implant.

SECONDARY OUTCOMES:
Crown contour of the tested implant | At least 12 months following implant placement.
  It is a one-time measurement (this study is only one-time visit) within the study timeframe. It is measured on ultrasound images. It is the angle between the tangent line of the implant crown and implant fixture.

CONTACTS AND LOCATIONS:
Overall Officials: Hsun-Liang Chan, DDS, MS, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan School of Dentistry
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abduo J. Axial Tooth Contour Alteration Following Fixed Prosthodontic Treatment. Eur J Prosthodont Restor Dent. 2014 Dec;22(4):174-82. PMID 26466442
- [Background] Berglundh T, Abrahamsson I, Welander M, Lang NP, Lindhe J. Morphogenesis of the peri-implant mucosa: an experimental study in dogs. Clin Oral Implants Res. 2007 Feb;18(1):1-8. doi: 10.1111/j.1600-0501.2006.01380.x. PMID 17224016
- [Background] Bichacho N, Landsberg CJ. Single implant restorations: prosthetically induced soft tissue topography. Pract Periodontics Aesthet Dent. 1997 Sep;9(7):745-52; quiz 754. PMID 9743681
- [Background] Canullo L, Tallarico M, Radovanovic S, Delibasic B, Covani U, Rakic M. Distinguishing predictive profiles for patient-based risk assessment and diagnostics of plaque induced, surgically and prosthetically triggered peri-implantitis. Clin Oral Implants Res. 2016 Oct;27(10):1243-1250. doi: 10.1111/clr.12738. Epub 2015 Nov 20. PMID 26584716
- [Background] Chan HL, Garaicoa-Pazmino C, Suarez F, Monje A, Benavides E, Oh TJ, Wang HL. Incidence of implant buccal plate fenestration in the esthetic zone: a cone beam computed tomography study. Int J Oral Maxillofac Implants. 2014 Jan-Feb;29(1):171-7. doi: 10.11607/jomi.3397. PMID 24451868
- [Background] Chan HL, Sinjab K, Chung MP, Chiang YC, Wang HL, Giannobile WV, Kripfgans OD. Non-invasive evaluation of facial crestal bone with ultrasonography. PLoS One. 2017 Feb 8;12(2):e0171237. doi: 10.1371/journal.pone.0171237. eCollection 2017. PMID 28178323
- [Background] Chan HL, Wang HL, Fowlkes JB, Giannobile WV, Kripfgans OD. Non-ionizing real-time ultrasonography in implant and oral surgery: A feasibility study. Clin Oral Implants Res. 2017 Mar;28(3):341-347. doi: 10.1111/clr.12805. Epub 2016 Mar 19. PMID 26992276
- [Background] Chifor R, Hedesiu M, Bolfa P, Catoi C, Crisan M, Serbanescu A, Badea AF, Moga I, Badea ME. The evaluation of 20 MHz ultrasonography, computed tomography scans as compared to direct microscopy for periodontal system assessment. Med Ultrason. 2011 Jun;13(2):120-6. PMID 21655538
- [Background] Chu SJ, Paravina RD. Periodontal-prosthodontics in contemporary practice. J Dent. 2013 Aug;41 Suppl 3:e1-2. doi: 10.1016/j.jdent.2013.06.010. No abstract available. PMID 23856512
- [Background] Cooper LF, Pin-Harry OC. "Rules of Six"--diagnostic and therapeutic guidelines for single-tooth implant success. Compend Contin Educ Dent. 2013 Feb;34(2):94-8, 100-1; quiz 102, 117. PMID 23556318
- [Background] Davarpanah M, Martinez H, Tecucianu JF. Apical-coronal implant position: recent surgical proposals. Technical note. Int J Oral Maxillofac Implants. 2000 Nov-Dec;15(6):865-72. PMID 11151587
- [Background] De Bruyckere T, Eghbali A, Younes F, De Bruyn H, Cosyn J. Horizontal stability of connective tissue grafts at the buccal aspect of single implants: a 1-year prospective case series. J Clin Periodontol. 2015 Sep;42(9):876-882. doi: 10.1111/jcpe.12448. Epub 2015 Sep 16. PMID 26373422
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Dierens M, de Bruecker E, Vandeweghe S, Kisch J, de Bruyn H, Cosyn J. Alterations in soft tissue levels and aesthetics over a 16-22 year period following single implant treatment in periodontally-healthy patients: a retrospective case series. J Clin Periodontol. 2013 Mar;40(3):311-8. doi: 10.1111/jcpe.12049. Epub 2013 Jan 9. PMID 23297745
- [Background] Du JK, Li HY, Wu JH, Lee HE, Wang CH. Emergence angles of the cementoenamel junction in natural maxillary anterior teeth. J Esthet Restor Dent. 2011 Dec;23(6):362-9. doi: 10.1111/j.1708-8240.2011.00471.x. Epub 2011 Sep 20. PMID 22142293
- [Background] Eghbali A, De Bruyn H, Cosyn J, Kerckaert I, Van Hoof T. Ultrasonic Assessment of Mucosal Thickness around Implants: Validity, Reproducibility, and Stability of Connective Tissue Grafts at the Buccal Aspect. Clin Implant Dent Relat Res. 2016 Feb;18(1):51-61. doi: 10.1111/cid.12245. Epub 2014 Jul 17. PMID 25040828
- [Background] Ericsson I, Lindhe J. Probing depth at implants and teeth. An experimental study in the dog. J Clin Periodontol. 1993 Oct;20(9):623-7. doi: 10.1111/j.1600-051x.1993.tb00706.x. PMID 8227448
- [Background] Funato A, Salama MA, Ishikawa T, Garber DA, Salama H. Timing, positioning, and sequential staging in esthetic implant therapy: a four-dimensional perspective. Int J Periodontics Restorative Dent. 2007 Aug;27(4):313-23. PMID 17726987
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Garber DA, Belser UC. Restoration-driven implant placement with restoration-generated site development. Compend Contin Educ Dent. 1995 Aug;16(8):796, 798-802, 804. PMID 8620398
- [Background] Grunder U, Gracis S, Capelli M. Influence of the 3-D bone-to-implant relationship on esthetics. Int J Periodontics Restorative Dent. 2005 Apr;25(2):113-9. PMID 15839587
- [Background] Ishikawa T, Salama M, Funato A, Kitajima H, Moroi H, Salama H, Garber D. Three-dimensional bone and soft tissue requirements for optimizing esthetic results in compromised cases with multiple implants. Int J Periodontics Restorative Dent. 2010 Oct;30(5):503-11. PMID 20814604
- [Background] Katafuchi M, Weinstein BF, Leroux BG, Chen YW, Daubert DM. Restoration contour is a risk indicator for peri-implantitis: A cross-sectional radiographic analysis. J Clin Periodontol. 2018 Feb;45(2):225-232. doi: 10.1111/jcpe.12829. Epub 2017 Dec 5. PMID 28985447
- [Background] Kois JC. Predictable single tooth peri-implant esthetics: five diagnostic keys. Compend Contin Educ Dent. 2001 Mar;22(3):199-206; quiz 208. PMID 11913257
- [Background] Le BT, Borzabadi-Farahani A, Pluemsakunthai W. Is buccolingual angulation of maxillary anterior implants associated with the crestal labial soft tissue thickness? Int J Oral Maxillofac Surg. 2014 Jul;43(7):874-8. doi: 10.1016/j.ijom.2014.02.009. Epub 2014 Mar 15. PMID 24637160
- [Background] Lee EA. Transitional custom abutments: optimizing aesthetic treatment in implant-supported restorations. Pract Periodontics Aesthet Dent. 1999 Nov-Dec;11(9):1027-34; quiz 1036. PMID 10853587
- [Background] Lin GH, Chan HL, Wang HL. Effects of currently available surgical and restorative interventions on reducing midfacial mucosal recession of immediately placed single-tooth implants: a systematic review. J Periodontol. 2014 Jan;85(1):92-102. doi: 10.1902/jop.2013.130064. Epub 2013 Apr 11. PMID 23578250
- [Background] Linkevicius T, Vindasiute E, Puisys A, Peciuliene V. The influence of margin location on the amount of undetected cement excess after delivery of cement-retained implant restorations. Clin Oral Implants Res. 2011 Dec;22(12):1379-84. doi: 10.1111/j.1600-0501.2010.02119.x. Epub 2011 Mar 8. PMID 21382089
- [Background] Listgarten MA, Lang NP, Schroeder HE, Schroeder A. Periodontal tissues and their counterparts around endosseous implants [corrected and republished with original paging, article orginally printed in Clin Oral Implants Res 1991 Jan-Mar;2(1):1-19]. Clin Oral Implants Res. 1991 Jul-Sep;2(3):1-19. doi: 10.1034/j.1600-0501.1991.020309.x. No abstract available. PMID 1843462
- [Background] Muller HP, Barrieshi-Nusair KM, Kononen E. Repeatability of ultrasonic determination of gingival thickness. Clin Oral Investig. 2007 Dec;11(4):439-42. doi: 10.1007/s00784-007-0125-0. Epub 2007 May 24. PMID 17522899
- [Background] Muller HP, Schaller N, Eger T. Ultrasonic determination of thickness of masticatory mucosa: a methodologic study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Aug;88(2):248-53. doi: 10.1016/s1079-2104(99)70123-x. PMID 10468471
- [Background] Nguyen KC, Le LH, Kaipatur NR, Major PW. Imaging the Cemento-Enamel Junction Using a 20-MHz Ultrasonic Transducer. Ultrasound Med Biol. 2016 Jan;42(1):333-8. doi: 10.1016/j.ultrasmedbio.2015.09.012. Epub 2015 Nov 3. PMID 26546266
- [Background] Nguyen KT, Le LH, Kaipatur NR, Zheng R, Lou EH, Major PW. High-Resolution Ultrasonic Imaging of Dento-Periodontal Tissues Using a Multi-Element Phased Array System. Ann Biomed Eng. 2016 Oct;44(10):2874-2886. doi: 10.1007/s10439-016-1634-2. Epub 2016 May 9. PMID 27160674
- [Background] Palou ME, McQuade MJ, Rossmann JA. The use of ultrasound for the determination of periodontal bone morphology. J Periodontol. 1987 Apr;58(4):262-5. doi: 10.1902/jop.1987.58.4.262. PMID 3295184
- [Background] Rompen E, Raepsaet N, Domken O, Touati B, Van Dooren E. Soft tissue stability at the facial aspect of gingivally converging abutments in the esthetic zone: a pilot clinical study. J Prosthet Dent. 2007 Jun;97(6 Suppl):S119-25. doi: 10.1016/S0022-3913(07)60015-8. PMID 17618926
- [Background] Saker S, El-Shahat S, Ghazy M. Fracture Resistance of Straight and Angulated Zirconia Implant Abutments Supporting Anterior Three-Unit Lithium Disilicate Fixed Dental Prostheses. Int J Oral Maxillofac Implants. 2016 Nov/Dec;31(6):1240-1246. doi: 10.11607/jomi.4131. PMID 27861648
- [Background] Scutella F, Weinstein T, Lazzara R, Testori T. Buccolingual implant position and vertical abutment finish line geometry: two strictly related factors that may influence the implant esthetic outcome. Implant Dent. 2015 Jun;24(3):343-8. doi: 10.1097/ID.0000000000000235. PMID 25764481
- [Background] Smukler H, Castellucci F, Capri D. The role of the implant housing in obtaining aesthetics: generation of peri-implant gingivae and papillae--Part 1. Pract Proced Aesthet Dent. 2003 Mar;15(2):141-9; quiz 150. PMID 12772631
- [Background] Spray JR, Black CG, Morris HF, Ochi S. The influence of bone thickness on facial marginal bone response: stage 1 placement through stage 2 uncovering. Ann Periodontol. 2000 Dec;5(1):119-28. doi: 10.1902/annals.2000.5.1.119. PMID 11885170
- [Background] Steigmann M, Monje A, Chan HL, Wang HL. Emergence profile design based on implant position in the esthetic zone. Int J Periodontics Restorative Dent. 2014 Jul-Aug;34(4):559-63. doi: 10.11607/prd.2016. PMID 25006773
- [Background] Su H, Gonzalez-Martin O, Weisgold A, Lee E. Considerations of implant abutment and crown contour: critical contour and subcritical contour. Int J Periodontics Restorative Dent. 2010 Aug;30(4):335-43. PMID 20664835
- [Background] Thoma DS, Sanz Martin I, Benic GI, Roos M, Hammerle CH. Prospective randomized controlled clinical study comparing two dental implant systems: demographic and radiographic results at one year of loading. Clin Oral Implants Res. 2014 Feb;25(2):142-9. doi: 10.1111/clr.12120. Epub 2013 Feb 19. PMID 23418746
- [Background] Tsiolis FI, Needleman IG, Griffiths GS. Periodontal ultrasonography. J Clin Periodontol. 2003 Oct;30(10):849-54. doi: 10.1034/j.1600-051x.2003.00380.x. PMID 14710764
- [Background] Tzoumpas M, Mohr B, Kurtulus-Waschulewski I, Wahl G. The Use of High-Frequency Ultrasound in the Measurement of Thickness of the Maxillary Attached Gingiva. Int J Prosthodont. 2015 Jul-Aug;28(4):374-82. doi: 10.11607/ijp.4250. PMID 26218020